CLINICAL TRIAL: NCT03975634
Title: Transcutaneous Spinal Stimulation: Augmenting Training for Attaining Intrinsic Trunk Control in Children With Spinal Cord Injury
Brief Title: Transcutaneous Spinal Stimulation: Safety and Feasibility for Trunk Control in Children With Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Andrea L. Behrman, PhD, PT, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19.0377
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: pediatric-onset; transcutaneous spinal stimulation; trunk control
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous spinal stimulation (Experimental): Safety and feasibility outcome measures are collected during application of transcutaneous spinal stimulation while trunk control is assessed at 3 time points (acute) and/or while transcutaneous stimulation is applied in combination with activity-based locomotor training (40 sessions, 1.5 hours/day, 5 days/week; stimulation will be applied intermittently for no more than 10 minutes at a time during training)
  Interventions: Device: Transcutaneous Spinal Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Stimulation — Safety and feasibility will be monitored during transcutaneous spinal stimulation in children with spinal cord injury

SUMMARY:
Paralysis of trunk muscles and the inability to sit upright is one of the major problems facing adults and children with spinal cord injury (SCI). Activity-based locomotor training has resulted in improved trunk control in children with spinal cord injury, though full recovery is not achieved in all children. Transcutaneous spinal stimulation' (TcStim), a stimulation applied over the skin to the sensory nerves and spinal cord, is a promising tool that may further enhance improvements to trunk control. The purpose of this study is to determine the feasibility (can we do it) and safety of Transcutaneous Stimulation (TcStim) in children with SCI to acutely improve sitting upright and when used with activity-based locomotor training (AB-LT). Thus, can we provide this therapy to children and do so safely examining a child's immediate response and cumulative response relative to safety and comfort.

Eight participants in this study will sit as best they can with and without the stimulation (i.e. stimulation applied across the skin to the nerves entering the spinal cord and to the spinal cord) and their immediate response (safety, comfort, trunk position) recorded. Then, two participants will receive approximately 40 sessions of activity-based locomotor training in combination with the stimulation. Their cumulative response of stimulation (i.e. safety, comfort, feasibility) across time will be documented. Participation in this study may last up to 3 days for the 8 participants being observed for acute response to stimulation and up to 9 weeks for the participants being observed for cumulative response to training with stimulation. We will monitor the participants throughout the testing and training for their response to the stimulation (i.e. safety) and their comfort.

DETAILED DESCRIPTION:
Similar to adults, children with severe spinal cord injury (SCI) suffer the devastating consequences of limb and trunk muscle paralysis rendering them unable to sit upright, stand, or walk. Unique to pediatric-onset SCI, nearly 100% of children injured under the age of 10 develop neuromuscular scoliosis with approximately 65% requiring surgical intervention. Given the importance of muscle activity and load-bearing for musculoskeletal development, SCI-induced trunk muscle paralysis during rapid growth contributes significantly to the onset and progression of scoliosis. Current physical rehabilitation interventions after pediatric-onset SCI are based on the premise of permanence of SCI-induced paralysis and the inability to restore intrinsic trunk control. As a result, thoraco-lumbosacral braces remain the standard of care for upright sitting support without clear efficacy for reducing the incidence of neuromuscular scoliosis.

Advances in rehabilitation after SCI, for adult and pediatric populations, capitalize on the intrinsic capacity of spinal neuronal networks for generation of motor output below the lesion in response to sensory input during activity-based locomotor training (AB-LT). Our recent work demonstrated remarkable improvements in trunk control as measured by the Segmental Assessment of Trunk Control (SATCo) in all 21 participants with SCI, age range: 17 months-12 years at enrollment and mean time since injury 1.5 years (range 1 month-6 years), receiving AB-LT across 60 sessions. Sensory-afferent driven activation of the intrinsic synergies between the lower limb and trunk extensor muscles above, across and below the lesion likely underlies the physiological adaptations responsible for these gains. While all children improved, not all attained full trunk control. Incorporation of neuromodulatory techniques, such as epidural spinal cord stimulation, further challenges the limits for SCI recovery previously thought possible. There are recent reports of individuals with chronic complete SCI regaining the capacity to stand and walk with stimulation. Transcutaneous spinal stimulation (TcStim) provides a non-invasive neuromodulatory tool that may, similar to epidural stimulation, increase the central state of excitability below the lesion, thereby enabling greater capacity for integration of sensory input and augment motor output to potentiate trunk motor recovery. Children with SCI may not only benefit from novel neurotherapeutic interventions, but also may demonstrate even greater improvements due to inherent plasticity present during development. Previous studies demonstrated the efficacy of TcStim to acutely improve sitting posture and trunk muscle activation in adults with SCI. In children with cerebral palsy, TcStim combined with AB-LT significantly improved locomotion compared to AB-LT alone. Our overall objective is to demonstrate 'proof-of-principle', as a necessary first step, that TcStim is a feasible and safe approach to a therapeutic intervention targeting trunk control in children with SCI. If found to be feasible and safe, then future studies will employ TcStim in combination with restorative rehabilitation for children with SCI to examine the effect on trunk control.

ELIGIBILITY:
Inclusion Criteria:

* history of chronic, acquired upper motor neuron SCI (traumatic or non-traumatic);
* discharged from in-patient rehabilitation
* moderate to severe trunk control deficit as either documented with the Segmental Assessment of Trunk Control (SATCo, score < 15/20) or reported/observed inability to sit fully upright and without use of arm support
* history of completion of a minimum of 60 sessions of activity-based locomotor training/therapy at Frazier Rehab

Exclusion Criteria:

* botox use within past 3 months;
* current baclofen use
* unhealed fracture
* any other medical complication limiting participation in the assessments and/or activity-based locomotor training;
* prior surgery for scoliosis;
* congenital SCI
* total ventilator dependence

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of skin irritation | 1 week for Aim 1, 9 weeks for Aim 2
  Skin color, particularly change in skin color to pink indicating irritation in the location of the stimulating electrode placement will be assessed prior to stimulation experiments and immediately after; incidence of pink- or redness or irritation and time (minutes-days) to dissipation will be recorded.
Faces Pain Scale-Revised (scale 0-10) | 1 week for Aim 1, 9 weeks for Aim 2
  Faces Pain Scale - Revised is a self-report measure of pain intensity developed for children (C.L. Hicks et al. Pain 93 (2001). It will be used to score the sensation of pain on 0 (min - no pain)-to-10 (max - worst pain ever) metric. The scale depicts 6 facial expressions: first - face with a neutral expression corresponds to pain score of 0, next facial expression is scored as 2, etc. The faces scale will be presented to the participant (ages 3-8) prior to the experiment for baseline measurement, during stimulation and following the experiment.
Visual Analog Scale (0-10) | 1 week for Aim 1, 9 weeks for Aim 2
  To assess pain in the participants ages 8 and above, Visual Analog Scale (self-reported measure) will be presented with 0 corresponding to no pain and 10 corresponding to the "worst pain ever"; the scale will be presented at baseline measurement, during stimulation and following the experiment.
Blood pressure | 1 week for Aim 1, 9 weeks for Aim 2
  continuous beat-by-beat blood pressure (mmHg) recordings will be made using Finapress finger cuff system for 5 minutes prior to and 5 minutes immediately following stimulation while the child is sitting; Brachial arm blood pressure will be periodically measured during stimulation (mmHg).
  systolic and diastolic blood pressure values will be compared with the established norms for typically developing children (age and height matched);
number of requests to stop the stimulation | 1 week for Aim 1, 9 weeks for Aim 2
  Number of participants requesting (or number of request per participant within experimental sessions) to stop stimulation due to pain, fatigue or any other reason (documented)
Angular excursions of trunk during trunk control assessments | 3 days for Aim 1, 9 weeks for Aim 2
  trunk kinematics (degrees of flexion/extension) in cervical, thoracic and lumbar regions;

SECONDARY OUTCOMES:
Heart rate | 1 week for Aim 1, 9 weeks for Aim 2
  heart rate (beats per minute) will be continuously monitored and recorded using 3-lead ECG electrocardiogram.
  The slope and correlation coefficient between beat-by-beat blood pressure and R-R intervals (ms) (measured from ECG) for 5 minutes prior to and 5 minutes immediately following stimulation will be used to assess spontaneous baroreflex sensitivity, indication of autonomic regulation of the cardiovascular function
Compliance rate | 1 week for Aim 1, 9 weeks for Aim 2
  Compliance - number of sessions missed and reason, willingness to continue participation.
Center of pressure displacement during trunk control assessment | 1 week for Aim 1, 9 weeks for Aim 2
  the distance (mm) of the center of pressure displacement will be measured in mediolateral; anterior -posterior directions during reaching tasks while the participant is sitting on the force plate

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PhD, PT, Principal Investigator — University of Louisville
Locations (1):
- Kentucky Spinal Cord Injury Res Center, University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keller A, Singh G, Sommerfeld JH, King M, Parikh P, Ugiliweneza B, D'Amico J, Gerasimenko Y, Behrman AL. Noninvasive spinal stimulation safely enables upright posture in children with spinal cord injury. Nat Commun. 2021 Oct 6;12(1):5850. doi: 10.1038/s41467-021-26026-z. PMID 34615867